CLINICAL TRIAL: NCT00506714
Title: Walking Aids in the Management of Hip Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arthritis Foundation (Other)
Responsible Party: Principal Investigator, Meika A. Fang, MD, Rheumatology, Arthritis Foundation
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007-030430
Record Dates: First submitted 2007-07-20; First posted 2007-07-25 (Estimated); Results first posted 2012-09-28 (Estimated); Last update posted 2012-10-04 (Estimated); Status verified 2012-09

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis; Walking Sticks; Canes
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adult subjects with hip osteoarthritis (Experimental): Walk with and without a single point cane at baseline and after four weeks
  Interventions: Device: single point cane
- Healthy Subjects (No Intervention): Healthy adults walking without a cane at baseline

INTERVENTIONS:
Device: single point cane — Adjustable single point cane with SureGrip handle
  Arms: Adult subjects with hip osteoarthritis

SUMMARY:
The purpose of this study is to determine whether or not the use of a nonpharmacologic intervention (single point cane) is effective in the treatment of knee osteoarthritis.

DETAILED DESCRIPTION:
Osteoarthritis (OA), the most common joint disease in humans, is a significant cause of pain and disability. Non-pharmacological treatments for hip OA include education, exercise, appliances (walking sticks or insoles), and weight reduction if obese or overweight. Canes are often recommended to reduce adverse forces across joints although there is currently no research evidence regarding the efficacy of walking sticks for hip OA. Little information is available regarding the impact of walking aids on psychosocial function and quality of life in individuals with hip OA. This study will evaluate the effects of walking aids in hip OA by examining gait biomechanics, quality of life, pain, and opinions regarding using a cane.

Comparisons: Compare gait biomechanics in people with symptomatic unilateral hip OA while walking with and without a cane at baseline and after 4 weeks of cane use. Compare gait biomechanics in people with symptomatic unilateral hip OA with and without a cane to those of healthy, age-matched controls. Compare pain and health-related quality of life in people with symptomatic unilateral hip OA following 4 weeks of cane use. Determine the association between changes in gait biomechanics, pain, and health-related quality of life in people with symptomatic unilateral hip OA following 4 weeks of cane use.

ELIGIBILITY:
Inclusion Criteria:

1. hip OA (grades II-IV) of the Kellgren/Lawrence classification
2. with pain in one hip for most days of the prior month
3. Ability to walk 30 feet without postural sway
4. Ability to stand unaided
5. Ability to understand verbal instructions
6. Ability to give informed consent

Exclusion Criteria:

1. History of hip or knee trauma or surgery including arthroscopic surgery in the past six months
2. Severe obesity (> 300 pounds)
3. Neurological disorders that affect lower extremity function such as stroke or peripheral neuropathy, vestibular dysfunction or poor vision
4. Injury or amputation to the lower extremity joints
5. History of other types of arthritis or fibromyalgia
6. Pain from spine, knee, ankle, or foot disease that would interfere with assessment of the hip
7. Poor health that would impair compliance or assessment such as shortness of breath with exertion, chest pain
8. Foot deformities such as hallux rigidus, valgus deformity of the midfoot, previous ankle arthrodesis
9. Greater trochanteric pain syndrome

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2007-07; Primary Completion 2009-07 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meika A Fang, MD, Principal Investigator — VA Greater Los Angeles Healthcare System Department of Medicine; UCLA Department of Medicine
Locations (1):
- VA West Los Angeles, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Healthy adults
- Group 2: Adults with symptomatic hip osteoarthritis
Period: Overall Study
Arm/Group | Group 1 | Group 2
Started | 13 | 13
Completed | 13 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 5 | 11
  >=65 years | 7 | 8 | 15
Age Continuous [Mean (Standard Deviation); unit: years] | 65 (4.4) | 67 (5.9) | 66 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 11 | 11 | 22
Region of Enrollment [Number; unit: participants]
  United States | 13 | 13 | 26

OUTCOME MEASURES:

1. Primary Outcome: Gait Velocity
Time Frame: Baseline
Population: Analysis was per protocol
Measure: Mean (Standard Deviation); unit: cm/s
Groups:
- Group 1: Healthy adults walking without a cane at baseline
- Group 2: Adults with symptomatic hip osteoarthritis walking without a cane at baseline
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 13 | 13
cm/s | 107.5 (14.3) | 79.7 (9.9)

2. Secondary Outcome: Gait Velocity With a Cane in Hip OA Subjects
Description: Measured gait velocity when hip OA subjects walked with a cane at the baseline visit.
Time Frame: Baseline
Population: Analysis was per protocol
Measure: Mean (Standard Deviation); unit: cm/s
Groups:
- Group 2: Adults with symptomatic hip osteoarthritis walking with a cane at baseline
Arm/Group | Group 2
Number analyzed (Participants) | 13
cm/s | 68.7 (15.4)

3. Secondary Outcome: Gait Velocity
Description: Gait velocity when adults with symptomatic hip osteoarthritis walked with a cane after four weeks of cane use
Time Frame: 4 weeks
Population: Analysis was per protocol
Measure: Mean (Standard Deviation); unit: cm/s
Groups:
- Group 2: Adults with symptomatic hip osteoarthritis after four weeks of cane use
Arm/Group | Group 2
Number analyzed (Participants) | 13
cm/s | 74.5 (14.2)

ADVERSE EVENTS:
Arm/Group | Group 1 | Group 2
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No